CLINICAL TRIAL: NCT04333836
Title: Comparison of the Efficiency of Maxillary Canine Retraction Using Aligners Versus Conventional Brackets in Orthodontic Extraction Cases.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Mostafa Osman Ramadan, Principle Inestigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aligners in Canine Retraction
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Removable Aligners, Conventional Brackets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aligners group (Experimental): Receiving full set of aligners ( Clear Removable Orthodontic appliance) until complete canine retraction
  Interventions: Device: Removable Clear Aligners
- Conventional Brackets group (Active Comparator): leveling and alignment of lower followed by complete canine retraction
  Interventions: Device: Removable Clear Aligners

INTERVENTIONS:
Device: Removable Clear Aligners — 1. Plaster dental models will be poured from the rubber base impression.
  2. Digital dental models will be created through scanning of plaster dental models.
  3. Planning of the aligners will be done on 3 shape clear aligner studio®.
  4. Aligners will be fabricated on 3d printed models using vacuum formers.
  5. Anchorage reinforcement for posterior segments by using buccal miniscrews.
  6. Patient will receive the first aligner and will be instructed to wear it full time (except during eating and brushing) for 2 weeks.
  7. Patient will receive the following aligner after 2 weeks.
  8. Follow up visits every 2 weeks until complete canine retraction.

SUMMARY:
The aim of this study is to compare the effectiveness of Clear aligners and Conventional braces for upper canine retraction (space closure) regarding canine tipping , anchorage loss and treatment time.

DETAILED DESCRIPTION:
Conventional fixed orthodontic treatment with metal brackets has been rejected by some adult patients because of esthetic and social concerns, but the demand for orthodontic treatment is currently increasing. To satisfy the demands and needs of these patients, the emphasis has shifted toward esthetic orthodontic appliance system. Less noticeable appliances such as ceramic, resin, and lingual brackets, or removable clear appliances such as the Essix and Invisalign (Align Technology, Santa Clara, Calif) provide esthetic orthodontic appliance alternatives.

Since the introduction of clear aligners to the public in 1999, it has become a popular treatment choice for clinicians because of the aesthetics and comfort of the removable clear aligners compared with traditional appliances. Several studies have shown significant limitations of this technique, especially in treating complex malocclusions, whereas other studies have reported successfully treated cases with this removable appliance. A systematic review conducted to determine the treatment effects of clear aligners showed that no strong conclusions could be made regarding the treatment effects of aligners . Therefore, clinical trials were still required to investigate the effectiveness of the Invisalign system.

When using the aligners to correct severe crowding, root positions must be carefully controlled during extraction space closure, and clear aligners must be properly grip all teeth to be moved, Tipping was a common problem in premolar extraction cases during the early years of aligners use. Several previous reports have also discussed the limited ability of thermoplastic appliances to control root-tipping movements and to establish root control comparable to that provided by fixed appliances. The investigators describe the extraction treatment of a patient with moderate to severe tooth crowding using mini screws and clear appliances, thus eliminating the need for conventional brackets.

ELIGIBILITY:
Inclusion Criteria:

* 1) Moderate to severe crowding orthodontic patients.( Irregularity index of <5 mm)

  2) Good oral hygiene. (Patient with periodontally sound dentition).

  3) Patient in permanent dentition between the age range 16 - 40 years.

  4) .Patients requiring extraction of mandibular and maxillary first premolars;

  5) Patients having sound general health

Exclusion Criteria:

* 1) Systematic disease.

  2) Poor oral hygiene patients.

  3 ) Periodontally affected teeth.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Canine Retraction (Space Closure ) | 6 months
  measured in millimeters

SECONDARY OUTCOMES:
Canine Tipping | 6 months
  it will be assessed by Angle degrees
Anchorage loss | 6 months
  it will be assessed by Angle degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Amr Mostafa Osman Ramadan, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided